CLINICAL TRIAL: NCT02467738
Title: A Pilot Study Using Surgical Resection and Intraoperative Cesium-131 Permanent Interstitial Brachytherapy Implant in Resectable Recurrent Head and Neck Cancer
Brief Title: Surgical Resection and Intraoperative Cesium-131 Brachytherapy for Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15D.067; 2014-112 (Other: CCRRC); JT 7243 (Other: JeffTrial Number)
Record Dates: First submitted 2015-06-05; First posted 2015-06-10 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Recurrent Head and Neck Carcinoma
MeSH Terms: interventions — Brachytherapy; Cesium-131

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cesium-131 Brachytherapy (Experimental): Patients undergo brachytherapy using Cesium-131 during surgical resection
  Interventions: Radiation: Brachytherapy; Drug: Cesium-131; Procedure: Conventional surgery

INTERVENTIONS:
Radiation: Brachytherapy — Undergo brachytherapy with Cesium-131
Drug: Cesium-131 — Undergo brachytherapy with Cesium-131
Procedure: Conventional surgery — Undergo surgical resection

SUMMARY:
This pilot clinical trial studies cesium Cs 131 brachytherapy in treating patients with head and neck cancer that has come back (recurrent) and can be removed by surgery. Brachytherapy, also known as internal radiation therapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. Radioactive drugs, such as cesium Cs 131, may carry radiation directly to tumor cells and not harm normal cells. Permanently implanting cesium Cs 131 into the wound bed after surgery may help treat microscopic cancer cells that may be in the tissue after surgical removal of the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the impact of cesium 131 (cesium Cs 131) on recurrence rate, disease free survival and over all survival.

SECONDARY OBJECTIVES:

I. Assess complications associated with cesium 131 treatment in subjects with head and neck cancer.

OUTLINE:

Patients undergo brachytherapy using cesium Cs 131 during surgical resection.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: Subjects with a diagnosis of recurrent head and neck cancer
2. Based on clinical and radiographic evidence the tumor needs to be deemed resectable preoperatively
3. Age: Subjects must be ≥ 18 years of age and ≤ 90 years old
4. Informed Consent: All subjects must be able to comprehend and sign a written informed consent document

Exclusion Criteria:

1. Subjects who are pregnant or may become pregnant
2. Unresectable tumor
3. Other severe acute or chronic medical or psychiatric condition that may increase the risk associated with study participation, and in the judgment of the investigator would make the subject inappropriate for entry into this study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2020-05-28 (Actual)

PRIMARY OUTCOMES:
Disease free survival (DFS) | Up to 24 months
  Will assess the impact of cesium Cs 131 on DFS by comparing the cohort to a matched historical control cohort. The distribution of DFS will be estimated using the Kaplan-Meier and a stratified log rank test will be used to test for differences between cohorts. Adjustment for other potential confounders will be performed using stratified Cox proportional hazards regression
Incidence of toxicity | Up to 90 days
  Evaluated using the Radiation Therapy Oncology Group Common Toxicity Criteria
  Categories of risk include infection, wound breakdown, inability to heal, fistula formation, bleeding and need for further surgery.

SECONDARY OUTCOMES:
Recurrence rate | Up to 24 months
  Comparisons of 6-month and one-year recurrence rates will be performed using logistic regression
Overall survival | Up to 24 months
  The distribution of overall survival will be estimated using the Kaplan-Meier and a stratified log rank test will be used to test for differences between cohorts. Adjustment for other potential confounders will be performed using stratified Cox proportional hazards regression.
Complication rate | Up to 24 months
  Estimated by cohort along with exact 95% confidence intervals
Adverse event rate | Up to 30 days
  Evaluated using the National Cancer Institute, Common Terminology Criteria for Adverse Events version 4.0
  Estimated by cohort along with exact 95% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Adam Luginbuhl, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Luginbuhl A, Calder A, Kutler D, Zender C, Wise-Draper T, Patel J, Cheng M, Karivedu V, Zhan T, Parashar B, Gulati S, Yao M, Lavertu P, Takiar V, Tang A, Johnson J, Keane W, Curry J, Cognetti D, Bar-Ad V. Multi-Institutional Study Validates Safety of Intraoperative Cesium-131 Brachytherapy for Treatment of Recurrent Head and Neck Cancer. Front Oncol. 2021 Nov 26;11:786216. doi: 10.3389/fonc.2021.786216. eCollection 2021. PMID 34900741
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/